CLINICAL TRIAL: NCT06315348
Title: Effect on the Periodontal Phenotype of Flapless Alveolar Decortication and Augmentation During Orthodontic Treatment: A Randomized Clinical Trial
Brief Title: Effect on Periodontal Phenotype of Flapless Piezoincission During Orthodontic Treatment
Acronym: Piezo_Ortho
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URI_116301123
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Dental Malocclusion; Maxillary Deficiency
Keywords: Periodontal phenotype; Flapless piezoincision; Orthodontic tooth movement; Tissue augmentation
MeSH Terms: conditions — Malocclusion; Retrognathia

STUDY DESIGN:
Intervention Model Description: Comparative 2-arm parallel double-blinded randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded parties will not be aware of the type augmentation used during the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen matrix (Experimental): a cross-linked volume stable collagen matrix (VCMX; Geistlich Fibro-Gide, Geistlich Pharma AG)
  Interventions: Procedure: flapless alveolar decortication with augmentation
- Xenograft (Active Comparator): a graft consisting of bovine hydroxyapatite xenograft (Geistlich Bio-Oss; Geistlich Pharma AG), covered by a native collagen membrane (Geistlich Bio-Gide; Geistlich Pharma AG), tagged with pins at the ends.
  Interventions: Procedure: flapless alveolar decortication with augmentation

INTERVENTIONS:
Procedure: flapless alveolar decortication with augmentation — piezocision-assisted orthodontics, concomitant to soft tissue grafting (volume-stable collagen matrix), with piezocision-assisted orthodontics, concomitant to bone grafting with a xenograft and a native collagen membrane. Piezocisions will be performed using a piezoelectric device.
  Other Names: flapless piezoincision with augmentation

SUMMARY:
Research Question

While the reduction in treatment times and the patient satisfaction after periodontally accelerated osteogenic orthodontics (PAOO) are well sustained in the scientific literature, there is still controversy regarding if grafting leads to i) change of the periodontal phenotype and ii) greater stability of post-orthodontic treatment outcomes, highlighting the need of controlled clinical trials.

Aims of the Project

The aim of this randomized clinical trial (RCT) is to compare piezocision-assisted orthodontics, concomitant to soft tissue grafting (volume-stable collagen matrix), with piezocision-assisted orthodontics, concomitant to bone grafting with a xenograft and a native collagen membrane, in orthodontic non-growing patients. The primary aim will be to determine the impact of this surgical protocol on the hard and soft tissue changes occurring on the buccal aspect of the dentition. Secondary objectives will include the assessment of the comparative impact on treatment duration, rate of tooth movements, presence of root resorption, periodontal parameters, bone level changes and patient-reported outcome measures (PROMs) between the two groups.

DETAILED DESCRIPTION:
Methodology

Study Design and Population Sample The study is designed as a single-blind (examiner), parallel groups, RCT to compare piezocision-assisted orthodontics concomitant to soft tissue grafting (soft tissue thickening group) or to bone grafting (bone augmentation group).

Patient Inclusion: Informed Consent, Patient Registration and Randomization If a patient fulfills the described inclusion/exclusion criteria, he/she will be invited to join the study. After informing the patient about the objectives, interventions, risks, benefits, and monitoring of the study, they will be asked to sign an informed consent form. Both the protocol of the study and consent forms have been approved by the local ethics committee at Hospital Clínico San Carlos (internal code 23/463-E, August 29, 2023).

Study Visits - Baseline Pretreatment orthodontic analysis will consist on intraoral scanner, panoramic x-rays, lateral cephalograms, CBCT scan and extra- and intra-oral photographs. Full-mouth periodontal examinations, including measurements of probing depth (PD) and gingival recession/overgrowth, will be taken at six sites per tooth, in all teeth excluding third molars, and will be rounded to the nearest millimetre using a UNC-15 probe. Plaque index (PlI) and bleeding on probing (BoP) will be also registered. The thickness of the soft tissue will be measured by an ultrasound scanner (PIROP Biometric G-Scan, Echoson Company, Poland), while the microvascularization will be measured by Laser Speckle Contrast Imaging (LSCI, PeriCam PSI System; Perimed AB, Sweden).

Study Visits - Orthodontic Treatment Orthodontic treatment will be carried out with clear or metal brackets (patients will be allowed to choose). The bonding method will be standardized and applied according to the manufacturer's instructions. After bracket bonding, 0.012-in. nickel-titanium arches forms will be placed. Subjects will return every other week and the archwires will be changed only when full bracket engagement will be achieved. The sequence of archwires will be as follows: 0.018-in., 0.014 × 0.025-in., and 0.018 × 0.025-in. copper nickel-titanium archwires were used for alignment, while 0.019 × 0.025-in. stainless-steel archwires were used for fine-tuning. Following the alignment steps, impressions will be taken, and a blinded senior orthodontist will validate appliance removal or provided advice regarding further adjustments. The study will end six months after the piezoincisions, when it is expected that a square or rectangular stainless-steel arch will be placed.

Study Visits - Surgical Procedures Piezocision surgical procedures will be performed one week after the placement of the orthodontic appliances (passive braces only, without arch-wires). After local anesthesia, vertical releasing incisions will be created at the distal aspect of the region to augment. Full thickness flaps will be raised and with a piezoelectric device, approximately 3 mm deep corticotomies will be made in between the dental roots. In case of root proximity (i.e. <2 mm of interdental bone), this procedure will not be performed. Then patients will be randomized to receive either i) a cross-linked volume stable collagen matrix (VCMX; Geistlich Fibro-Gide, Geistlich Pharma AG); or ii) a graft consisting of bovine hydroxyapatite xenograft (Geistlich Bio-Oss; Geistlich Pharma AG) that will be covered by a native collagen membrane (Geistlich Bio-Gide; Geistlich Pharma AG), tagged with pins at the ends.

Finally, resorbable sutures will be used in the microincisions. The microvasculature and the thickness of the soft tissue will be measured right after the surgery on the same measurement areas. The patients will be advised to take analgesics only if necessary and to record their daily intake for one week. Anti-inflammatories will be prohibited to avoid interference with the RAP. Careful brushing and the use of a 0.12% chlorhexidine mouthwash will be recommended for 7 days after surgery.

Immediately after surgery, the arch-wires will be placed and orthodontic tooth movement will start.

Study Visits - Follow-up Following the alignment steps, intraoral scanners will be taken every month during the first 6 months, and a blinded orthodontist will validate appliance removal or provide advice for further adjustments. At 6 months and at the time of removal of appliances, a new intraoral scanner will be taken, and a full-mouth periodontal chart performed. The measurement of microvasculature and soft tissue thickness will be executed at the same region of interests. Patients will be monitored regarding their periodontal status throughout the study. Patients presenting ≥2 sites with attachment loss ≥2 mm or FMPS ≥ 25% will be exited from the study.

Superimposed STL files will allow for measuring the changes in tissue contours and buccal volume. Furthermore, the superimposition of STL and DICOM files will allow to evaluate changes in buccal bone and soft tissue thickness (i.e. periodontal phenotype). Space analyses, including intercanine and intermolar distances, as well as upper and lower central incisor angles, will be performed at baseline and after the end of the treatment on the STL files with digital tools. Times from bracket placement to removal will be recorded in days.

Outcome Variables - Periodontal Outcomes:

Clinical periodontal parameters will be recorded at six sites per tooth, in all teeth excluding third molars, at the beginning and at the end (6 months?) of the orthodontic therapy:

* PlI will be dichotomously assessed and expressed as the percentage of positive sites out of the total sites assessed.
* BOP will be dichotomously assessed and expressed as the percentage of positive sites out of the total sites assessed.
* PD and gingival recession/overgrowth, allowing for the calculation of clinical attachment level (CAL).

Outcome Variables - Orthodontic Parameters:

Space analyses will be performed on study models with digital calipers. Similarly, the intercanine and intermolar distances will be measured at baseline and after the treatments to determine the level of expansion. The upper and lower central incisor angles will be calculated according to lateral cephalometric x-rays. The cumulative times from bracket placement to each archwire change and to orthodontic appliance removal will be recorded in number of days.

Outcome Variables - Primary outcomes based on image analysis:

The study casts will be optically scanned with a desktop 3D scanner (Zfx Evolution Scanner, Zimmer Dental. Bolzano, Italy). The baseline and post-ortho STL files will be uploaded to an image analysis software (SMOP, Swissmeda Ltd©, Zurich, Switzerland). For matching the STL files, three clear and visible pairs of reference points will be selected in both the baseline and follow-up casts allowing the software to perform a "rough fit." After this, additional references (no fewer than 10) will be selected to assist the matching and perform a "fine fit" of the surfaces. Then using a series of mathematical algorithms to achieve a "best-fit," the software automatically will superimpose the models.

The superimposed STL file allows for measuring the changes in tissue contour pre- and post- orthodontic therapy:

1. Linear measurements: from the cross-sectional views at the middle of the crown of selected teeth at baseline, a line coinciding with the axis of the tooth was drawn and then, perpendicular lines to this axis were drawn at 1, 2, 3, 4, and 5 below the gingival margin (GM). The horizontal dimensions of the tissue contours were then measured at these different heights at baseline and after orthodontic treatment. Also, the gingival recession was assessed by measuring the distance of GM at the different time points.
2. Volumetric measurements: a selected area of interest delimited by the gingival margin around selected teeth, and by the mesial and distal line angles extending 5-6 mm apically will be drawn to evaluate the volume changes. The software will calculate a value corresponding to the mean distance in millimeters between the two surface areas, and then the volume change in cubic millimeters corresponding to the volume enclosed between the two surfaces.
3. Presence of root resorption (CBCT)

Outcome Variables - Secondary and explanatory outcomes:

The following will be considered:

* Percentage of residual pockets (PD>4 mm).
* Changes in soft tissue thickness by PIROP ultrasound scanner
* Changes in microvasculature by Laser Speckle Contrast Imaging before and after the surgical intervention
* PROMs, including impact on quality of life (GOHAI), pain level after treatment and daily analgesic consumption following piezoincisions (questionnaires will be provided at 72 h and d15 days). After the overall treatment, the levels of satisfaction in terms of the final result, the treatment duration, and whether the patient would recommend the procedure to a friend will be assessed. Finally, the patients were asked whether they would undergo the treatment again.
* Presence of adverse events (AEs).

Data Analyses and Sample Size Calculation:

Sample size calculation was performed for the primary outcome variable, changes in buccal bone and soft tissue thickness, considering a standard deviation of 0.8 mm and a desirable difference between groups of 1 mm, with a 90% of power, resulting in a sample of 14 patients per arm. To compensate for dropouts, a desired number of 20 patients per arm will be aimed.

The normality of the distribution will be assessed; evaluating skewness, kurtosis, and using the Kolmogorov-Smirnov test. ANOVA and the multiple rank test will be used to compare the baseline visit with the 3- and 6-month visits (intra-group comparisons). ANCOVA will be used to compare both groups, at baseline or in changes baseline - follow-up visits (inter-group comparison); using treatment group as the factor and including baseline values of the examined variable, smoking and gender as cofactors. The level of statistical significance will be set at p≤0.05. However, because multiple comparisons will be carried out for the inter-group assessment, the Bonferroni correction will be used.

ELIGIBILITY:
Inclusion Criteria:

Patients will be consecutively selected among those attending the Faculty of Odontology, University Complutense (Madrid, Spain) looking for orthodontic therapy.

The inclusion criteria will be as follows:

* patients requiring maxillary and/or mandible orthodontic treatment;
* patients with permanent dentition in stage 5 or 6 of the cervical vertebral maturation method as described by Baccetti et al. (2002);
* minimal to moderate maxillary and/or mandibular anterior crowding at baseline (arch length discrepancy from 3-8 mm); and
* adequate oral health (i.e. periodontal health, absence of periapical infections and untreated caries).

Exclusion Criteria:

* subjects with periodontitis stage III or IV (Papapanou et al., 2018);
* subjects with poor oral hygiene (represented as full-mouth plaque scores (FMPS) >25%);
* ongoing chronic drug therapy influencing bone metabolism (e.g. steroids, immunosuppressors or antiresorptive drugs);
* subjects with uncontrolled systemic diseases (e.g. diabetes);
* pregnancy and
* subjects not willing to comply with the study visits

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Soft tissue contour changes pre- and post- orthodontic therapy | 6 months
  Linear and volumetric changes of soft tissue (gingiva) using superimposition of STL files of dental casts at baseline and post-ortho
Plaque index (PlI) | 6 months
  Changes in PlI dichotomously assessed and expressed as the percentage of positive sites out of the total sites assessed.
Bleeding on probbing (BoP) | 6 months
  Changes in BoP dichotomously assessed and expressed as the percentage of positive sites out of the total sites assessed
Probing depth (PD) | 6 months
  Changes in PD and gingival recession/overgrowth, allowing for the calculation of clinical attachment level (CAL)
External apical root resorption (EARR) | 6 months
  Presence of EARR measured in 3D Cone bean computed tomography (CBCT)
Orthodontic tooth movement | 6 months
  Space analyses will be performed on study models with digital calipers. Similarly, the intercanine and intermolar distances will be measured at baseline and after the treatment to determine the level of expansion

SECONDARY OUTCOMES:
Percentage of residual pockets (PD>4 mm). | 6 months
  Percentage of residual pockets (PD>4 mm).
Soft tissue thickness by PIROP ultrasound scanner | 6 months
  Changes in soft tissue thickness by PIROP ultrasound scanner
Gingival microvasculature | 6 months
  Changes in microvasculature by Laser Speckle Contrast Imaging before and after the surgical intervention
PROMs | 72 h and 15 days
  PROMs including impact on quality of life (GOHAI), pain level after treatment and daily analgesic consumption following piezoincisions
Adverse events (AEs) | During the study duration (6 months)
  Presence of adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Odontology, University Complutense Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request

REFERENCES:
- [Result] REFERENCE LIST Charavet, C., Lecloux, G., Bruwier, A., Rompen, E., Maes, N., Limme, M., & Lambert, F. (2016). Localized Piezoelectric Alveolar Decortication for Orthodontic Treatment in Adults: A Randomized Controlled Trial. J Dent Res, 95(9), 1003-1009. doi:10.1177/0022034516645066 Charavet, C., Lecloux, G., Jackers, N., Albert, A., & Lambert, F. (2019). Piezocision-assisted orthodontic treatment using CAD/CAM customized orthodontic appliances: a randomized controlled trial in adults. Eur J Orthod, 41(5), 495-501. doi:10.1093/ejo/cjy082 Charavet, C., Lecloux, G., Jackers, N., Maes, N., & Lambert, F. (2019). Patient-reported outcomes measures (PROMs) following a piezocision-assisted versus conventional orthodontic treatments: a randomized controlled trial in adults. Clin Oral Investig, 23(12), 4355-4363. doi:10.1007/s00784-019-02887-z